CLINICAL TRIAL: NCT05023733
Title: Clinical and Radiographic Outcomes of Transforaminal Lumbar Interbody Fusion (TLIF) With a Novel 3D Printed Cellular Titanium Implant
Brief Title: Clinical and Radiographic Outcomes of TLIF w/3D Printed Cellular Implant
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Farhan Karim (Other)
Collaborators: DePuy Synthes (Industry)
Responsible Party: Sponsor-Investigator, Farhan Karim, Spine Surgeon, Hartford Hospital
Organization: Hartford Hospital (Other)
Other Study IDs: HHC-2020-0243
Record Dates: First submitted 2021-08-16; First posted 2021-08-27 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Foraminal Stenosis; Degenerative Disc Disease; Lumbar Spondylolisthesis; Lumbar Spinal Stenosis
Keywords: transforaminal; degenerative disc disease (DDD); Lumbar Fusion; Interbody Fusion
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spondylolisthesis; Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- 1-2 contiguous levels of interbody fixation from a transforaminal approach for spinal segments L2-S1: One to two contiguous levels of interbody fixation from a transforaminal approach for spinal segments L2-S1 whose condition requires the use of interbody fusion.
  Interventions: Device: CONDUIT™ Interbody Platform composed of the EIT (Emerging Implant Technologies) Cellular Titanium®

INTERVENTIONS:
Device: CONDUIT™ Interbody Platform composed of the EIT (Emerging Implant Technologies) Cellular Titanium® — Patients undergoing 1-2 contiguous levels of interbody fixation from a transforaminal approach for spinal segments L2-S1
  Other Names: lumbar fusion

SUMMARY:
This study is designed to evaluate clinical outcomes and spine fusion rates for patients undergoing transforaminal lumbar interbody fusion using the CONDUIT 3D printed titanium TLIF cage.

DETAILED DESCRIPTION:
This prospective, single-center study is being conducted as a post market evaluation of the CONDUIT 3D printed titanium TLIF Cage. Patients undergoing transforaminal lumbar interbody fusions due to lumbar spinal pathology (i.e. central foraminal stenosis, degenerative disc disease, and/or lumbar spondylolisthesis) and have failed conservative care will be recruited for this study. Patients will be serially evaluated at 6 month intervals for a total of 24 months post index procedure to assess patient reported outcomes, clinical outcomes, and radiographic parameter, specifically spine fusion rates.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature adults ages 35 - 80 years of age, inclusive
* Diagnosis of lumbar degenerative disc disease with or without neurologic deficit and associated central and/or unilateral/bilateral foraminal stenosis
* Subject undergoing one or two level transforaminal lumbar interbody fusion
* Able to read and understand all documents used in this study , including the informed consent and patient-reported outcome questionnaires

Exclusion Criteria:

* Patients over 80 years of age
* Patients under 35 years of age
* Current smokers
* BMI>42
* Subject has spondylolisthesis > 2
* Subjects with multilevel >2 levels of symptomatic disease
* Subjects with significant spinal deformity
* Subject is pregnant, plans to become pregnant or is breast feeding

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be skeletally mature adults ages 35-80 years of age undergoing one or two level transforaminal lumbar interbody fusion. These patients will have a diagnosis of lumbar degenerative disc disease with or without neurologic deficit and associated central and/or unilateral /bilateral foraminal stenosis.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Radiographic Fusion | 18 months
  Fusion success measured by radiological assessment. Evidence of fusion demonstrated by bone formation through the cage on anteroposterior (AP) and Lateral radiographs, Flexion and Extension radiographs at 18 months
Radiographic Fusion | 24 months
  Fusion success measured by radiological assessment. Evidence of fusion demonstrated by bone formation through the cage on anteroposterior (AP) and Lateral radiographs, Flexion and Extension radiographs at 24 months

SECONDARY OUTCOMES:
Back and Leg Visual Analog Scale (VAS) | 6 months
  Improvement in the VAS as measured by a minimum of a 20 point improvement
Back and Leg Visual Analog Scale (VAS) | 12 months
  Improvement in the VAS as measured by a minimum of a 20 point improvement
Back and Leg Visual Analog Scale | 18 months
  Improvement in the VAS as measured by a minimum of a 20 point improvement
Oswestry Disability Index (ODI) | 6 months
  Clinical Improvement will be defined by improvement in Oswestry Disability Index (ODI) >20%
Oswestry Disability Index (ODI) | 12 months
  Clinical Improvement will be defined by improvement in Oswestry Disability Index (ODI) >20%
Oswestry Disability Index (ODI) | 18 months
  Clinical Improvement will be defined by improvement in Oswestry Disability Index (ODI) >20%
Adverse Events | up to 24 months
  Number of procedure and device related adverse events
Intervention Rates | up to 24 months
  Rates of reoperation and/or revision procedures at index level(s)

CONTACTS AND LOCATIONS:
Overall Officials: Farhan Karim, DO, Principal Investigator — Hartford Hospital; Hartford Healthcare Bone & Joint Institute
Locations (1):
- Hartford Healthcare Bone and Joint Institute, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided